CLINICAL TRIAL: NCT04931069
Title: Correlation Between Complications After Pancreaticoduodenectomy and Biliary, Pancreatic, Blood, Oral, Intestinal and Fecal Microbiota
Brief Title: Correlation Between Complications After Pancreaticoduodenectomy and Microbiota
Acronym: COMPAMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/21/0004
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
Keywords: microbiota; microbiome; pancreaticoduodenectomy; pancreatic resection; Whipple procedure; postoperative complications
MeSH Terms: conditions — Pancreatic Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Microbiota analysis (Experimental): Mircobiota analysis on blood, stool and saliva and bile, pancreatic and intestinal mucosa samples
  Interventions: Other: Microbiota analysis

INTERVENTIONS:
Other: Microbiota analysis — Microbiota analysis will be carried out on different samples: blood, stool and saliva samples will be collected during the surgery, between 5 and 10 days after surgery and at 3 and 6 months after the surgery. Bile, pancreatic and intestinal mucosa samples will only be collected during the surgery.

SUMMARY:
Pancreaticoduodenectomy is the most performed pancreatic surgery for malignant or premalignant tumors of the region of the head of the pancreas. Its post-operative morbidity is very high, over 40%. There is very little data on the impact of microbiota on complications after pancreatic surgery. The purpose of this research is to study the correlation between the microbiota (fecal, blood, oral, biliary, pancreatic and intestinal microbiota) and the postoperative complications in patients who undergo pancreaticoduodenectomy.

DETAILED DESCRIPTION:
After pancreaticoduodenectomy, the post-operative complications can be surgical (pancreatic fistula, gastroparesis) but also infectious, digestive (diarrhea) and lead to malnutrition. They are responsible for prolonged post-operative hospitalizations, impaired quality of life of patients and induce a delay in the implementation of adjuvant chemotherapy, or even an impossibility to achieve it. The absence of adjuvant chemotherapy adversely affects the prognosis of patients, by increasing the rate of recurrence and decreased survival. There is therefore a real oncological benefit in finding solutions to reduce the number and severity of these complications. A change in post-operative microbiota composition has been shown to play a role in the development of post-surgical anastomotic fistulas in colorectal cancer. Despite their importance, there is very little data on the impact of microbiota on complications after pancreatic surgery. We postulate that microbiota variations could have an impact on early and late post-operative complications after pancreaticoduodenectomy. Any patient hospitalized at the Toulouse University Hospital with an indication of a pancreaticoduodenectomy will be offered to participate in this study. Microbiota analysis will be carried out on different samples: blood, stool and saliva samples will be collected during the surgery, between J5 and J10 (post-operative during hospitalization) and at 3 and 6 months after the surgery. Bile, pancreatic and intestinal mucosa samples will only be collected during the surgery. Complications will be collected throughout this study. This study will not create any additional constraints on patient management. The follow-up period will be 6 months. This follow-up period will be fixed for all patients included. The microbiota analyses will be centrally determined during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized at the Toulouse University Hospital with an indication of a pancreaticoduodenectomy
* Patient aged over 18 years old
* Patient having given his written consent
* Patient with social insurance coverage

Exclusion Criteria:

* Patient for whom the pancreaticoduodenectomy was not realized (exploratory laparotomy or other surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Analysis of the microbiota | within 90 days after surgery
  the analysis of the microbiota on the per-operative samples (fecal, blood, oral, biliary, pancreatic and intestinal) in patients undergoing pancreaticoduodenectomy according to the occurrence of early post-operative complications (≤ 90 days)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte MAULAT, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No